CLINICAL TRIAL: NCT04201509
Title: Validity of Neurocognitive Assessment Methods in Childhood ADHD
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/88
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Neurodevelopmental Disorders; Attention Deficit Hyperactivity Disorder
Keywords: Intelligence; Anxiety; Attention; Conduct behavior; Follow-up; Children
MeSH Terms: conditions — Neurodevelopmental Disorders; Attention Deficit Disorder with Hyperactivity; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADHD group: Participants in the clinical group were recruited to the project when they were assessed for and diagnosed with ADHD at the Neuropsychiatric Unit of the CAP Clinic in Lund in 2011-2012. The ADHD group was treated as usual in the clinic and re-assessed during 2014-2015.
- Non-clinical group: Participants in the non-clinical group were recruited recruited 2012 from schools in the same district and among children of the same average age as the ADHD-group 2012. The non-clinical group did not have any intervention during the follow-up time. Th non-clinical group was re-assessed during 2015.

SUMMARY:
The aim of the study is to examine the prospective validity of neurocognitive functions and emotional factors in schoolchildren with ADHD and a control group of typically developing schoolchildren at baseline and after three years.

DETAILED DESCRIPTION:
In spite of extensive research on children with ADHD, there is still insufficient understanding of the discriminative validity of neurocognitive tests and how test results of neurocognitive functions and ratings of emotional factors and ADHD symptoms change over time and interacts during development. The project is studying the validity of clinical assessment methods within the Swedish child and adolescent psychiatry service (CAP) related to the identification of ADHD, additional impairments, and comorbidity. The prospective validity of neurocognitive functions and emotional factors in schoolchildren with ADHD and a control group of typically developing schoolchildren at baseline and after three years will be investigated.

Specific aims: Aim I: Study how attentiveness and impulsivity in ADHD change over three years by comparing the results of psychological tests and rating scales at baseline and after three years Aim II: Study intellectual development in ADHD by comparing the results of intelligence tests at baseline and after three years- Aim III: Study how emotional factors change over three years by comparing the results of rating scales at baseline and after three years

ELIGIBILITY:
Inclusion Criteria: The ADHD-group:

• The individuals were assessed and diagnosed with ADHD at the Neuropsychiatric Unit of the CAP Clinic in Lund in 2011-2012

Non-clinical group:

* School children from Lund.

Exclusion Criteria:

* If the individual had a diagnosed intellectual disability
* If the individual required an interpreter to participate in the study

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children diagnosed with ADHD at the Neuropsychiatric Unit of the CAP Clinic in Lund in 2011-2012, 7 to 18 years old when recrutited to the study. School children from Lund, 7 to 18 years old when recrutited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Emotional status assessed with the Beck Youth Inventory. | 2011-2012 and 2014-2015
  The children were assessed with the Beck youth scales at two timepoints with a time interval of 3 years. Beck Youth Inventory consist of 5 subscales, Depression, Anxiety, Anger, Disruptive behaviour, Self-concept. It is standardized into percentiles and higher scores mean worse behaviour, except for Self-concept. In Self-concept higher scores mean better behaviour.

SECONDARY OUTCOMES:
Neuropsychological status assesses with the Conners' Continuous Performance Test (CPT) II | 2011-2012 and 2014-2015
  The children were assessed with the Conners'CPT II at two timepoints with a time interval of 3 years. Conners' CPT II is a performance based test measuring reaction time, reaction time variability, omissions and comissions. Conners' CPT II is standardised into T scores; mean=50, SD=10. Higher scores mean worse results.

OTHER OUTCOMES:
Cognitive status assesses with the Weschsler Intelligence Scales for Children-Fourth Edition (WISC-IV) | 2011-2012 and 2014-2015
  The children were assessed with the WISC-IV at two timepoints with a time interval of 3 years. The WISC-IV is a performance based test, measuring cognitive functioning. The WISC-IV consists of 10 core subtests, that form four composites (Verbal Comprehension, Perceptual Reasoning, Working Memory, Processing Speed) and Full Scale IQ. The WISC-IV is standardised into the IQ scale, mean=100, SD=15. Higher scores mean better results.

CONTACTS AND LOCATIONS:
Overall Officials: Peik Gustafsson, Dr, Principal Investigator — Lund University
Locations (1):
- Pia Tallberg, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No